CLINICAL TRIAL: NCT04621097
Title: Effect of Pulsed Electrmagnetic Field Versus Treadmill Training on Walking and Haemodynamic Parameters in Peripheral Arterial Disease
Brief Title: Pulsed Electromagnetic Field Versus Treadmill Walking in Peripheral Arterial Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, reham raafat mahmoud, REHAM RAAFAT, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002122
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: group A : Pulsed electromagnetic field PLUS medications group B : Treadmill Training Plus Medications group C :medications only
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pulsed electro magnetic field (Experimental): 30 patients will receive the physical therapy program in form of low frequency pulsed electro magnetic field application. with frequency 15hz, and low intensity with flux density of 20 Gauss (2mT), in pulse duration 200 usec , pulsed rectangular pulses for 60 min is applied to the dorsal surface of lower leg , ankle and foot in addition to their regular medications prescribed , 3 times per week for 8 week
  Interventions: Device: pulsed electromagnetic field
- Treadmilltraining (Experimental): * In this group, 30 patient will receive the physical therapy program in form of supervised treadmill walking exercise. The exercise program consists of intermittent walking bouts to moderate claudication pain alternating with periods of rest in between for a total of 40-50 minutes .
  * At first , a 5 minutes- warm up period will be allowed, it will include stretching exercises for calf muscles , hamstrings and quadriceps (i.e. each for at least 10 -15 seconds) . Patients should start with walking on the treadmill at a comfortable speed, and should not stop at the onset of leg pain but instead , he/she would continue until moderate pain is reached. At this point, he/she has to rest until pain completely subsides, then walking is resumed again . The intensity of exercise will be determined by claudication pain scale, and should not exceed the score of 4 on this scale. The exercise can be progressed if the patient can walk continuously for 10 minutes without the need to stop.
  Interventions: Other: treadmill training
- medications (Placebo Comparator): It includes 20 patients who will not receive any physiotherapy intervention. They will receive medical treatment only and will act as a control group.
  Interventions: Drug: Medication

INTERVENTIONS:
Device: pulsed electromagnetic field — it is a device for magnetotherapy and it is one of the most recent noninvasive physical therapy modality which is used in multiple physical therapy fields . it consist of an appliance, motorized bed and solenoid . the appliance must be connected to electrical supplying 230 =10% at a frequency of 50 or 60 HZ with earth connection . the intensity and spatial lay out of the generated magnetic field depend on the type of solenoid used
  Other Names: BTL -5000 Magneto Therapy .
  Arms: pulsed electro magnetic field
Other: treadmill training — supervised treadmill walking exercise. The exercise program consists of intermittent walking bouts to moderate claudication pain alternating with periods of rest in between for a total of 40-50 minutes .
  Other Names: intermittent walking excercise
  Arms: Treadmilltraining
Drug: Medication — regular medications
  Arms: medications

SUMMARY:
my study is to determine the effect of pulsed electromagnetic field versus treadmill training in managemet of intemittent claudication in peripheral arterial disease

there is a lack of interventions that improves local peripheral blood circulation in ischemic lower limbs . (PEMFs) are a non-pharmacological and non-invasive treatment that can be applied on the affected body part, which penetrates through skin and reaches target tissues . However, there have been few clinical studies reporting the effects of PEMFs on hemodynamic response in people with PAD (

DETAILED DESCRIPTION:
Statement of the problem :

Is there any Difference between Pulsed ElectroMagnetic Field and Supervised Treadmill walking exercise on improving exercise performance and hemodynamic parameters in patients with peripheral arterial disease

The use of pulsed electromagnetic field (12hz to50hz) in improving microcirculation , microvascular blood perfusion , stimulation of nitric oxide release and stimulating angiogensis has introduced a new dimension to the physical therapy field , to the available knowledge puplished , there is no literature about analgesic and microcirculatory effect of PEMF on circulation improvement in patients with PAD , therefore the proplem of the study will be stated in a questionnary form for answering the following aspects : ( Chalidia B. etal 2011)

Significance of the study :

Treatment of PAD is critically important in order to minimize the risk of long term disability and improve quality of life . The need of this study developed from the lack in published studies about the effect of pulsed electromagnetic field in management of peripheral arterial diseases and also there was no available previous trials comparing the effect of PEMF and treadmill exercise on walking parameters , posterior tibial artery diameter and ABI on patients with PAD

the results of this study may provide an easy non pharmacological modality for dealing with such cases . Also, the outcome of this study will guide physiotherapists to develop a new noninvasive treatment modality that may improve patient symptoms and promotes their social participation , this in turn may add to clinical role played by therapists in management of intermittent claudication in patients with peripheral arterial diseases. In Addition, increased knowledge of the influence of PEMF on microvascular function may have significant therapeutic potential and may be valuable for the intervention of diabetes-related lower limb vascular occlusion and amputation in the clinic.

1. Does pulsed electromagnetic field will have an effect on posterior tibial artery diameter using Doppler ultrasound in patients with PAD and suffering from intermittent claudication ?
2. Does pulsed electromagnetic field will be effective in improving the claudication pain time and distance , maximal walking free time and distance in patients with peripheral arterial disease ?
3. Does pulsed electromagnetic field will be effective in improving the ABI ( ankle brachial pressure index in patients with peripheral arterial disease?
4. Does non invasive pulsed electromagnetic field (PEMF) will be better than supervised treadmill walking exercise in management of intermittent claudication in patients with peripheral arterial disease ?
5. Are there differences between PEMF and supervised treadmill walking exercise in improving exercise performance and hemodynamic parameters in patients with peripheral arterial diseases ?

Purpose of the study Purposes of this study will be the following

1. To evaluate the therapeutic efficacy of pulsed electromagnetic field On walking parameter (on Maximum walking Free time , Maximum walking Free distance, Claudication pain time , Claudication pain distance ) in management of intermittent claudication in patients with PAD .
2. To evaluate the effect of non invasive pulsed electromagnetic field on ABI (ankle brachial pressure index) in patients with PAD suffering from intermittent claudication.
3. To investigate the effect of non invasive PEMF on Posteriot Tibial Artery Diameter in patients with PAD suffering from intermittent claudication.
4. To evaluate the effect of supervised treadmill walking exercise in managemet of intermittent claudication in patients with PAD
5. to compare between the efficacy of non invasive pulsed electromagnetic field versus supervised treadmill walking exercise ( on distance and time till reaching maximum tolerated pain of intermittent claudication and also the efficacy on ankle brachial pressure index , pain intensity level ) in patients with peripheral arterial diseases suffering from intermittent claudication
6. To gain knowledge about Non Invasive Pulsed Electromagnetic Field application and implementation in physical therapy field
7. To share in designing an ideal protocol for the treatment of intermittent claudication in patients with PAD

ELIGIBILITY:
Inclusion Criteria:

* Both genders are allowed to participate in the study .
* The age range of patients will be from 45-65 years
* All patients are diagnosed with PAD since at least ( 6 months to1 year) and suffer from IC
* All patients will be suffering from moderate degree of pain in the calf according to claudication pain scale.
* ABPI for all patients will be ranged from 0.65 to 0. 9
* All patients are medically and psycholigically stable .
* Only ambulant patient without any aids will be selected
* All patients are non smokers

Exclusion Criteria:

* Patients with Severe grades of intermittent claudication that produce ischemic pain at rest
* Presence of claudication symptoms less than 2 months
* Patients with fontaine stage I PAD (asymptomatic)
* Patient with fontaine stage III PAD (leg pain at rest )
* Patients with ABPI ( Ankle Brachial Pressure Index ≤ 0.4 )
* Patients who are unable to walk on the treadmill or unable to attend sessions at the physical therapy department at APH , 3 times a week .
* Patients with unstable cardiovascular conditions (those with a known history of recent myocardial infarction, uncontrolled hypertension, ischemic attacks, stroke, congestive heart failure) will be excluded from this study.
* Patients with neurological problems that cause leg pain .
* Patients with active malignancy will be excluded from study Patients with acute tuberculosis, soft tissue infection, cellulities, hyperthyroidism, acute viral diseases, Patients with pace makers will be excluded from the study Patients with ischemic ulcers or gangrenes
* Patients with marked dyspnea on exertion or with chronic obstructive pulmonary diseases (COPD).
* Patients with a vascular surgical procedure or angioplasty within the previous year will be excluded from the study
* Patients with musculoskeletal disorders ( Diagnosed with severe osteoporosis , severe osteoarthritis or joint replacement )

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Ankle brachial pressure index ( ABPI ) | 8 weeks
  it will be measured by doppler ultrasound
Posterior Tibial Artery Diameter ( PTA ) | 8 WEEKS
  it will be measured by doppler ultrasound

SECONDARY OUTCOMES:
claudication onset time (COT) or distance | 8 WEEKS
  it will be measured by Graded Treadmill Exercise Testing
a peak walking time (PWT) or peak walking distance. | 8 WEEKS
  it will be measured by Graded treadmill exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: reham raafat, phd, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: within 6 months